CLINICAL TRIAL: NCT03648372
Title: An Open Label, Dose-Escalation, Phase 1/2 Study to Evaluate the Safety, Tolerability, Preliminary Efficacy and Pharmacokinetics of TAK-981 in Adult Patients With Advanced or Metastatic Solid Tumors or Relapsed/Refractory Hematologic Malignancies
Brief Title: A Study of TAK-981 in People With Advanced Solid Tumors or Cancers in the Immune System
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enrolment Challenges
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-981-1002; U1111-1214-4537 (Registry Identifier: WHO); 2020-003947-27 (EudraCT Number)
Record Dates: First submitted 2018-08-24; First posted 2018-08-27 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Neoplasms; Lymphoma; Hematologic Neoplasms
Keywords: Drug therapy
MeSH Terms: conditions — Neoplasms; Lymphoma; Hematologic Neoplasms | interventions — TAK-981

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase 1, Dose Escalation Cohort: TAK-981 (Experimental): TAK-981, intravenously, administered as 60 minute-infusion, once on Days 1, 4, 8, and 11 in a 21-day treatment cycle for up to approximately 12 months or until discontinuation from the study. If clinical safety, pharmacokinetics, and pharmacodynamics are supportive, the dosing schedule may be modified to evaluate a less intensive administration of TAK-981 on Day 1, or Days 1 and 8, or Day 1, Day 8, and Day 15 in 21-day cycles in participants with advanced or metastatic solid tumors or lymphomas. Dose levels will be escalated based on the Bayesian logistic regression modeling (BLRM). The dose escalation phase will determine the RP2D of TAK-981.
  Interventions: Drug: TAK-981
- Phase 2, Cohort A: Nonsquamous NSCLC (Experimental): TAK-981 intravenously administered as 60 minute-infusion in a 21-day treatment cycle for up to approximately 12 months or until discontinuation from the study in participants with nonsquamous non-small cell lung cancer (NSCLC).
  Interventions: Drug: TAK-981
- Phase 2, Cohort B: Cervical Cancer (Experimental): TAK-981 intravenously administered as 60 minute-infusion in a 21-day treatment cycle for up to approximately 12 months or until discontinuation from the study in participants with cervical cancer.
  Interventions: Drug: TAK-981
- Phase 2, Cohort C: MSS-CRC (Experimental): TAK-981 intravenously administered as 60 minute-infusion in a 21-day treatment cycle for up to approximately 12 months or until discontinuation from the study in participants with microsatellite-stable colorectal cancer (MSS-CRC).
  Interventions: Drug: TAK-981
- Phase 2, Cohort D: r/r DLBCL after CAR T-cells therapy (Experimental): TAK-981 intravenously administered as 60 minute-infusion in a 21-day treatment cycle for up to approximately 12 months or until discontinuation from the study in participants with relapsed/refractory (r/r) diffuse large B-cell lymphoma (DLBCL) after prior chimeric antigen receptor (CAR) T-cells therapy.
  Interventions: Drug: TAK-981
- Phase 2, Cohort E: r/r DLBCL without prior cellular therapy (Experimental): TAK-981 intravenously administered as 60 minute-infusion in a 21-day treatment cycle for up to approximately 12 months or until discontinuation from the study in participants with relapsed/refractory DLBCL that have not received prior cellular therapy.
  Interventions: Drug: TAK-981
- Phase 2, Cohort F: r/r Follicular Lymphoma (Experimental): TAK-981 intravenously administered as 60 minute-infusion in a 21-day treatment cycle for up to approximately 12 months or until discontinuation from the study in participants with relapsed/refractory follicular lymphoma (FL).
  Interventions: Drug: TAK-981

INTERVENTIONS:
Drug: TAK-981 — Intravenous infusion.

SUMMARY:
This study is in 2 parts.

The main aims of the 1st part of the study are to check if people with advanced solid tumors or cancers in the immune system (lymphomas) have side effects from TAK-981, and to check how much TAK-981 they can receive without getting side effects from it.

The main aims of the 2nd part of the study are to learn if the condition of people with specific cancers improves after treatment with TAK-981. Another aim is to check for side effects from TAK-981.

In the 1st part of the study, participants will receive TAK-981. In the 2nd part of the study, participants with specific tumor types will receive TAK-981 at the recommended phase 2 dose determined during the 1st part of the study.

In both parts of the study, participants can receive TAK-981 for up to 1 year or longer if their condition stays improved. Participants will receive TAK-981 through vein.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-981. TAK-981 is being tested to evaluate safety, tolerability, preliminary efficacy and PK in participants with advanced or metastatic solid tumors or relapsed/refractory hematologic malignancies. The study will include 2 phases: Phase 1 dose escalation and Phase 2 dose expansion cohorts (cancer treatment expansions).

The study will enrol approximately 202 participants, approximately 70 participants in the dose escalation phase, approximately 132 participants in cancer treatment expansion phase.

In the dose escalation, dose levels will be escalated based on safety, and available PK and pharmacodynamic data and will also determine the single agent RP2D. Participants in dose expansion phase will be enrolled, once RP2D is determined. There will be 6 cohorts in cancer treatment expansions.

* Cohort A: Nonsquamous NSCLC
* Cohort B: Cervical cancer
* Cohort C: MSS-CRC
* Cohort D: Relapsed/refractory DLBCL progressed or relapsed after CAR T-cells therapy
* Cohort E: Relapsed/refractory DLBCL that have not received prior cellular therapy
* Cohort F: Relapsed/refractory FL

This multi-center trial will be conducted in European Union, China and United States. The overall time to participate in this study is approximately 2 years. The overall time to receive treatment in the dose escalation and cancer treatment is approximately 1 year. Based on decision of sponsor, participants with demonstrated clinical benefit can continue treatment beyond 1 year. Participants will make multiple visits to the clinic and will make a final visit 30 days after receiving their last dose of drug or before the start of subsequent anticancer therapy, whichever occurs first for a follow-up assessment.uroped

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female participants ≥18 years old.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
3. Population for Phase 1 dose escalation:

   * Has histologically or cytologically confirmed advanced (local regionally recurrent not amenable to curative therapy) or metastatic solid tumors who have no standard therapeutic option with a proven clinical benefit, are intolerant, or have refused them. OR
   * Has relapsed/refractory lymphoma not amenable to therapies with proven clinical benefit or who are intolerant or who refuse them. Participants with low-grade lymphomas such as FL, small lymphocytic lymphoma, lymphoplasmacytoid lymphoma, and marginal zone lymphomas, may not need to exhaust all available therapy. These participants can be enrolled after failure of at least 2 prior systemic therapies, provided that there is not an immediate need for cytoreduction. In these cases, participants who need immediate therapy for tumor bulk are not eligible for this trial.
4. Population for Phase 2 dose expansion cohorts:

   o Has histologically or cytologically documented, advanced (metastatic and/or unresectable) cancer as listed below, that is incurable and for which prior standard first-line treatment has failed: Note: Prior neoadjuvant or adjuvant therapy included in initial treatment may not be considered first- or later-line SOC treatment unless such treatments were completed less than 12 months before the current tumor recurrence.

   o Nonsquamous NSCLC that has progressed to 1 prior systemic immune checkpoint inhibitors (CPI)/anti-PD-(1/L1)-containing therapy and no more than 2 lines of therapy. Participants must have not shown evidence of tumor progression during the first 5 months of treatment with first-line CPI/anti-PD-(1/L1)-containing therapy (cohort A).

   Note: Participants with known driver mutations/genomic aberrations (example- epidermal growth factor receptor [EGFR], B-Raf proto-oncogene mutation V600E [BRAF V600E], and ROS proto-oncogene 1 [ROS1] sensitizing mutations, neurotrophic receptor tyrosine kinase [NRTK] gene fusions, and anaplastic lymphoma kinase [ALK] rearrangements) must have also shown progressive disease after treatment with a commercially available targeted therapy.

   o CPI-naïve cervical cancer (squamous cell carcinoma, adenosquamous carcinoma or adenocarcinoma of the cervix) participants who have received no more than 1 prior systemic line of therapy for recurrent or Stage IVB cervical cancer (cohort B).

   Note: The following cervical tumors are not eligible: minimal deviation/adenoma malignum, gastric-type adenocarcinoma, clear-cell carcinoma, and mesonephric carcinoma. Histologic confirmation of the original primary tumor is required via pathology report.

   Note: First-line treatment must have consisted of platinum-containing doublet. Chemotherapy administered concurrently with primary radiation (example- weekly cisplatin) is not counted as a systemic chemotherapy regimen.

   o CPI-naïve MSS-CRC participants who have progressed on no more than 3 chemotherapy regimens (cohort C).

   Note: Participants must have received prior treatment with fluoropyrimidine-, oxaliplatin-, and irinotecan-containing regimens if indicated.
   * Relapsed/refractory DLBCL progressed or relapsed after prior CAR T cell therapy that has received approval by a health authority for the treatment of DLBCL (cohort D).
   * Relapsed/refractory DLBCL that has progressed or relapsed after at least 2 but no more than 3 prior lines of systemic therapy and has not received prior cellular therapy. At least one prior line of therapy must have included a CD20-targeted therapy (cohort E).
   * Relapsed/refractory FL that has progressed or relapsed after at least 2 but no more than 3 prior lines of systemic therapy. At least 1 prior line of therapy must have included a CD20-targeted therapy (cohort F).
5. In Phase 2 only, have at least 1 radiologically measurable lesion based on RECIST v1.1 for participants with solid tumors or Lugano criteria for lymphoma. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.

   Note: In Phase 2 stage 1, have an additional lesion for pretreatment and on-treatment biopsy.
6. In Phase 2 stage 1, willing to consent to mandatory pretreatment and on-treatment tumor biopsy.

   Note: For fresh tumor biopsies, the lesion must be accessible for a biopsy procedure as assessed by the investigator.
7. Is willing to provide archival tumor tissue sample, if available.
8. Adequate bone marrow reserve and renal and hepatic function.
9. Recovered to Grade 1 or baseline or established as sequelae from all toxic effects of previous therapy (except alopecia, neuropathy, or autoimmune endocrinopathies with stable endocrine replacement therapy, bone marrow parameters [any of Grade 1 or 2 permitted if directly related to bone marrow involvement).
10. Consented to undergo serial skin punch biopsies (dose escalation only).
11. Suitable venous access for safe drug administration and the study-required PK and pharmacodynamics sampling.
12. Women of childbearing potential participating in this study should avoid becoming pregnant, and male participants should avoid impregnating a female partner. Nonsterilized female participants of reproductive age and male participants should use effective methods of contraception through defined periods during and after study treatment as specified below. Female participants must meet 1 of the following:

    * Postmenopausal for at least 1 year before the screening visit, or
    * Surgically sterile, or
    * If they are of childbearing potential, agree to practice 1 highly effective method and 1 additional effective (barrier) method of contraception at the same time, from the time of signing of the informed consent form (ICF) through 6 months after the last dose of study drug, or
    * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [example, calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)
13. Male participants, even if surgically sterilized (that is, status post vasectomy) must agree to 1 of the following:

    * Agree to practice effective barrier contraception during the entire study treatment period and through 6 months after the last dose of study drug, or
    * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [example, calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)

Exclusion Criteria:

1. Phase 1 dose escalation and Phase 2 cancer treatment expansion cohorts:

   o Has received treatment with systemic anticancer treatments or investigational products within 14 days before the first dose of study drug or 5 half-lives, whichever is shorter.

   Note: Low-dose steroids (oral prednisone or equivalent ≤20 mg per day), hormonal therapy for prostate cancer or breast cancer (as adjuvant treatment), and treatment with bisphosphonates and receptor activator of nuclear factor kappa-Β ligand (RANKL) inhibitors are allowed.

   o Has received extended field radiotherapy ≤4 weeks before the start of treatment (≤2 weeks for limited field radiation for palliation), and who has not recovered to grade 1 or baseline from related side effects of such therapy (except for alopecia).
2. History of any of the following ≤6 months before first dose: congestive heart failure New York Heart Association Grade III or IV, unstable angina, myocardial infarction, unstable symptomatic ischemic heart disease, severe noncompensated hypertension despite appropriate medical therapy, ongoing symptomatic cardiac arrhythmias of >Grade 2, pulmonary embolism, or symptomatic cerebrovascular events, or any other serious cardiac condition (example, pericardial effusion or restrictive cardiomyopathy). Chronic atrial fibrillation on stable anticoagulant therapy is allowed.
3. Baseline prolongation of the QT interval with Fridericia correction method (QTcF) (example, repeated demonstration of QTcF interval >480 milliseconds (ms), history of congenital long QT syndrome, or torsades de pointes).
4. Psychiatric illness/social circumstances that would limit compliance with study requirements and substantially increase the risk of adverse events (AEs) or has compromised ability to provide written informed consent.
5. Admission or evidence of illicit drug use, drug abuse, or alcohol abuse.
6. History of autoimmune disease requiring systemic immunosuppressive therapy.
7. History of immune-related AEs related to treatment with immune checkpoint inhibitors that required treatment discontinuation.
8. History of noninfectious pneumonitis that required steroids or a history of interstitial lung disease.
9. Has evidence of active, noninfectious pneumonitis.
10. Have a significant active infection.
11. Known history of human immunodeficiency virus (HIV) infection or any other relevant congenital or acquired immunodeficiency.
12. Known hepatitis B virus (HBV) surface antigen seropositive or detectable hepatitis C infection viral load. Note: Participants who have positive hepatitis B core antibody or hepatitis B surface antigen antibody can be enrolled but must have an undetectable hepatitis B viral load.
13. Receiving or requiring the continued use of medications that are known to be strong or moderate inhibitors and inducers of cytochrome P-450 3A4/5 (CYP3A4/5) or are strong permeability glycoprotein (P-gp) inhibitors. To participate in this study, participants should discontinue use of such agents for at least 2 weeks (1 week for CYP3A4/5 and P-gp inhibitors) before receiving a dose of TAK-981.
14. Participant requires the use of drugs known to prolong QTc interval (during Phase 1 only).
15. History of allogeneic tissue or solid organ transplant.
16. Second malignancy within the previous 3 years, except treated basal cell or localized squamous skin carcinomas, localized prostate cancer, cervical carcinoma in situ, resected colorectal adenomatous polyps, breast cancer in situ, or other malignancy for which the participant is not on active anticancer therapy.
17. Female participants who are lactating and breastfeeding or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (8):
- United States (8):
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - HealthPartners Cancer Care Center - Regions Hospital, Saint Paul, Minnesota
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Nakamura A, Grossman S, Song K, Xega K, Zhang Y, Cvet D, Berger A, Shapiro G, Huszar D. The SUMOylation inhibitor subasumstat potentiates rituximab activity by IFN1-dependent macrophage and NK cell stimulation. Blood. 2022 May 5;139(18):2770-2781. doi: 10.1182/blood.2021014267. PMID 35226739
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b60354db2bf003ab4a092

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 17 investigative sites in Poland, Belgium, Spain, the United States and China from 01 October 2018 to 14 December 2023.
Pre-assignment Details: Participants were enrolled in Phase 1 (Dose Escalation) and in Phase 2 (Dose Expansion) to receive TAK-981 doses.
Groups:
- Phase 1, Dose Escalation: TAK-981 3 mg BIW: Participants with relapsed/refractory advanced or metastatic solid tumors or lymphoma received TAK-981 3 milligram (mg), infusion, intravenously, twice weekly (BIW) on Days 1, 4, 8 and 11 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 1, Dose Escalation: TAK-981 6 mg BIW: Participants with relapsed/refractory advanced or metastatic solid tumors or lymphoma received TAK-981 6 mg, infusion, intravenously, BIW on Days 1, 4, 8 and 11 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 1, Dose Escalation: TAK-981 10 mg BIW: Participants with relapsed/refractory advanced or metastatic solid tumors or lymphoma received TAK-981 10 mg, infusion, intravenously, BIW on Days 1, 4, 8 and 11 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 1, Dose Escalation: TAK-981 15 mg BIW: Participants with relapsed/refractory advanced or metastatic solid tumors or lymphoma received TAK-981 15 mg, infusion, intravenously, BIW on Days 1, 4, 8 and 11 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 1, Dose Escalation: TAK-981 25 mg BIW: Participants with relapsed/refractory advanced or metastatic solid tumors or lymphoma received TAK-981 25 mg, infusion, intravenously, BIW on Days 1, 4, 8 and 11 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 1, Dose Escalation: TAK-981 40 mg BIW: Participants with relapsed/refractory advanced or metastatic solid tumors or lymphoma received TAK-981 40 mg, infusion, intravenously, BIW on Days 1, 4, 8 and 11 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 1, Dose Escalation: TAK-981 60 mg BIW: Participants with relapsed/refractory advanced or metastatic solid tumors or lymphoma received TAK-981 60 mg, infusion, intravenously, BIW on Days 1, 4, 8 and 11 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 1, Dose Escalation: TAK-981 60 mg QW: Participants with relapsed/refractory advanced or metastatic solid tumors or lymphoma received TAK-981 60 mg, infusion, intravenously, once weekly (QW) on Days 1 and 8 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 1, Dose Escalation: TAK-981 75 mg BIW: Participants with relapsed/refractory advanced or metastatic solid tumors or lymphoma received TAK-981 75 mg, infusion, intravenously, BIW on Days 1, 4, 8 and 11 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 1, Dose Escalation: TAK-981 75 mg QW: Participants with relapsed/refractory advanced or metastatic solid tumors or lymphoma received TAK-981 75 mg, infusion, intravenously, QW on Days 1 and 8 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 1, Dose Escalation: TAK-981 90 mg BIW: Participants with relapsed/refractory advanced or metastatic solid tumors or lymphoma received TAK-981 90 mg, infusion, intravenously, BIW on Days 1, 4, 8 and 11 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 1, Dose Escalation: TAK-981 90 mg QW: Participants with relapsed/refractory advanced or metastatic solid tumors or lymphoma received TAK-981 90 mg, infusion, intravenously, QW on Days 1 and 8 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15: Participants with relapsed/refractory advanced or metastatic solid tumors or lymphoma received TAK-981 90 mg, infusion, intravenously, QW on Days 1, 8 and 15 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 1, Dose Escalation: TAK-981 120 mg BIW: Participants with relapsed/refractory advanced or metastatic solid tumors or lymphoma received TAK-981 120 mg, infusion, intravenously, BIW on Days 1, 4, 8 and 11 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 1, Dose Escalation: TAK-981 120 mg QW: Participants with relapsed/refractory advanced or metastatic solid tumors or lymphoma received TAK-981 120 mg, infusion, intravenously, QW on Days 1 and 8 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 2, Dose Expansion, Cohort A, NSCLC: TAK-981 90 mg BIW: Participants with non-squamous non-small cell lung cancer (NSCLC) received TAK-981 90 mg, infusion, intravenously, BIW on Days 1, 4, 8 and 11 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 2, Dose Expansion, Cohort B, Cervical Cancer: TAK-981 90 mg BIW: Participants with cervical cancer received TAK-981 90 mg, infusion, intravenously, BIW on Days 1, 4, 8 and 11 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 2, Dose Expansion, Cohort C, MSS-CRC: TAK-981 90 mg BIW: Participants with microsatellite-stable colorectal cancer (MSS-CRC) received TAK-981 90 mg, infusion, intravenously, BIW on Days 1, 4, 8 and 11 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 2, Dose Expansion, Cohort D, DLBCL After CAR T-cells Therapy: TAK-981 90 mg BIW: Participants with relapsed/refractory diffuse large B-cell lymphoma (DLBCL) progressed or relapsed after chimeric antigen receptor (CAR) T-cell therapy received TAK-981 90 mg, infusion, intravenously, BIW on Days 1, 4, 8 and 11 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 2, Dose Expansion, Cohort E, DLBCL Without Prior Cellular Therapy: TAK-981 90 mg BIW: Participants with relapsed/refractory DLBCL that have not received prior cellular therapy received TAK-981 90 mg, infusion, intravenously, BIW on Days 1, 4, 8 and 11 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 2, Dose Expansion, Cohort F, Follicular Lymphoma: TAK-981 90 mg BIW: Participants with relapsed/refractory follicular lymphoma received TAK-981 90 mg, infusion, intravenously, BIW on Days 1, 4, 8 and 11 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
Period: Overall Study
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW | Phase 2, Dose Expansion, Cohort A, NSCLC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort B, Cervical Cancer: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort C, MSS-CRC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort D, DLBCL After CAR T-cells Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort E, DLBCL Without Prior Cellular Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort F, Follicular Lymphoma: TAK-981 90 mg BIW
Started | 5 | 3 | 4 | 3 | 4 | 4 | 7 | 6 | 6 | 6 | 8 | 7 | 7 | 8 | 6 | 7 | 3 | 7 | 4 | 3 | 1
Completed | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 2 | 2 | 1 | 1 | 0 | 1 | 1 | 1 | 4 | 2 | 1
Not Completed | 4 | 3 | 4 | 3 | 3 | 3 | 5 | 5 | 5 | 5 | 6 | 5 | 6 | 7 | 6 | 6 | 2 | 6 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 2 | 3 | 4 | 3 | 2 | 2 | 3 | 3 | 5 | 5 | 2 | 3 | 3 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 3 | 0 | 5 | 1 | 5 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Start of a New Systemic Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set consisted of participants who received at least 1 dose, even if incomplete, of study drug.
Groups:
- Phase 1, Dose Escalation: TAK-981 3 mg BIW: Participants with relapsed/refractory advanced or metastatic solid tumors or lymphoma received TAK-981 3 mg, infusion, intravenously, BIW on Days 1, 4, 8 and 11 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Phase 1, Dose Escalation: TAK-981 60 mg QW: Participants with relapsed/refractory advanced or metastatic solid tumors or lymphoma received TAK-981 60 mg, infusion, intravenously, QW on Days 1 and 8 in a 21-day treatment cycle until confirmed disease progression, unacceptable toxicity, or any criterion for withdrawal from the study or discontinuation of study drug occurred.
- Total: Total of all reporting groups
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW | Phase 2, Dose Expansion, Cohort A, NSCLC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort B, Cervical Cancer: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort C, MSS-CRC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort D, DLBCL After CAR T-cells Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort E, DLBCL Without Prior Cellular Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort F, Follicular Lymphoma: TAK-981 90 mg BIW | Total
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 4 | 4 | 7 | 6 | 6 | 6 | 8 | 7 | 7 | 8 | 6 | 7 | 3 | 7 | 4 | 3 | 1 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (9.78) | 61.0 (14.73) | 52.0 (11.05) | 66.7 (10.69) | 59.5 (5.80) | 65.0 (4.69) | 59.3 (10.21) | 62.5 (9.07) | 60.8 (10.87) | 62.3 (10.97) | 60.5 (9.56) | 62.4 (14.21) | 64.4 (7.93) | 59.4 (11.02) | 57.8 (8.33) | 64.0 (6.98) | 53.3 (2.08) | 51.6 (13.02) | 56.3 (18.06) | 71.7 (5.51) | 53.0 (NA) — Standard Deviation could not be estimated due to insufficient number of participants available for analysis. | 60.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 4 | 4 | 3 | 5 | 4 | 3 | 5 | 1 | 3 | 3 | 0 | 3 | 1 | 58
  Male | 1 | 1 | 2 | 1 | 2 | 2 | 4 | 4 | 2 | 2 | 5 | 2 | 3 | 5 | 1 | 6 | 0 | 4 | 4 | 0 | 0 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 5 | 3 | 4 | 2 | 3 | 4 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 7 | 3 | 7 | 4 | 3 | 1 | 100
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 9
  White | 5 | 3 | 4 | 3 | 3 | 4 | 4 | 4 | 4 | 6 | 7 | 6 | 7 | 5 | 5 | 7 | 3 | 2 | 4 | 2 | 0 | 88
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants Reporting One or More Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs were adverse events (AEs) that occurred after administration of the first dose of any study drug and through 30 days after the last dose of any study drug. AE means any untoward medical occurrence in a participant administered a pharmaceutical product. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product. Any abnormal laboratory results were considered as TEAEs.
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (up to 35.3 months)
Population: Safety analysis set consisted of participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 4 | 4 | 7 | 6 | 6 | 6 | 8 | 7 | 7 | 8 | 6
Participants | 4 | 3 | 4 | 3 | 4 | 4 | 6 | 6 | 5 | 6 | 8 | 7 | 7 | 8 | 6

2. Primary Outcome: Phase 1: Number of Participants With Grade 3 or Higher TEAEs
Description: The severity grade was evaluated as per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0, except for Cytokine Release Syndrome (CRS), which was assessed by American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading. Where Grade 3 was severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living (ADL), Grade 4 was life-threatening consequences; urgent intervention indicated, and Grade 5 was death related to AE. TEAEs were AEs that occurred after administration of the first dose of any study drug and through 30 days after the last dose of any study drug.
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (up to 35.3 months)
Population: Safety analysis set consisted of participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 4 | 4 | 7 | 6 | 6 | 6 | 8 | 7 | 7 | 8 | 6
Participants | 2 | 2 | 3 | 1 | 2 | 2 | 4 | 3 | 4 | 0 | 6 | 5 | 4 | 7 | 3

3. Primary Outcome: Phase 1: Duration of TEAEs
Description: TEAEs were AEs that occurred after administration of the first dose of any study drug and through 30 days after the last dose of any study drug. AE means any untoward medical occurrence in a participant administered a pharmaceutical product. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product.
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (up to 35.3 months)
Population: Safety analysis set consisted of participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Median (Full Range); unit: days
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 4 | 4 | 7 | 6 | 6 | 6 | 8 | 7 | 7 | 8 | 6
days | 3.0 [1 to 37] | 4.0 [1 to 21] | 1.0 [1 to 33] | 3.0 [1 to 5] | 4.0 [1 to 39] | 9.5 [1 to 36] | 4.0 [1 to 42] | 3.0 [1 to 47] | 8.0 [1 to 82] | 2.0 [1 to 58] | 4.5 [1 to 188] | 5.0 [1 to 37] | 2.0 [1 to 80] | 3.0 [1 to 131] | 4.0 [1 to 64]

4. Primary Outcome: Phase 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs were evaluated according to NCI CTCAE version 5.0. Grade 5 AE. Hematologic toxicity: Nonfebrile Grade 4 neutropenia/Grade greater than or equal to (>=) 3 febrile neutropenia; Significant Grade 3 thrombocytopenia; Grade 4 thrombocytopenia. Nonhematologic Grade 3 or higher toxicities; Grade 2 nonhematologic toxicities that were considered by the investigator to be related to study drug and dose-limiting.
Time Frame: Cycle 1 (Cycle length is equal to [=] 21 days)
Population: DLT-evaluable analysis set consisted of participants in dose escalation who received all Cycle 1 doses of TAK-981 without experiencing a DLT or who had a DLT during Cycle 1 of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 4 | 4 | 6 | 5 | 5 | 6 | 6 | 6 | 7 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0

5. Primary Outcome: Phase 2: Overall Response Rate (ORR)
Description: ORR was defined as percentage of participants who achieved complete response (CR) or partial response (PR) during the study as determined by the investigator according to response assessments based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST V1.1) for solid tumors or Lugano classification for lymphoma.
Time Frame: From the first dose of study drug until first disease progression (PD) or death, whichever occurred first (up to 11.2 months)
Population: Tumor response-evaluable analysis set consisted of participants who received at least 1 dose of study drug, had sites of measurable disease at baseline, and 1 postbaseline disease assessment, or was discontinued due to symptomatic deterioration or death before a postbaseline evaluation happened.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2, Dose Expansion, Cohort A, NSCLC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort B, Cervical Cancer: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort C, MSS-CRC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort D, DLBCL After CAR T-cells Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort E, DLBCL Without Prior Cellular Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort F, Follicular Lymphoma: TAK-981 90 mg BIW
Number analyzed (Participants) | 7 | 3 | 6 | 4 | 3 | 1
percentage of participants | 0.0 [0.0 to 40.96] | 0.0 [0.0 to 70.76] | 0.0 [0.0 to 45.93] | 0.0 [0.0 to 60.24] | 0.0 [0.0 to 70.76] | 100.0 [2.50 to 100.0]

6. Secondary Outcome: Phase 1, Cmax: Maximum Observed Plasma Concentration for TAK-981
Description: Cmax for TAK-981 was reported.
Time Frame: Cycle 1 Day 1: pre-dose and at multiple timepoints (up to 48 hours) post-dose; Cycle 1 Day 8: pre-dose and at multiple timepoints (up to 24 hours) post-dose (Cycle length = 21 days)
Population: Pharmacokinetic (PK) analysis set consisted of participants with sufficient dosing and PK data to reliably estimate 1 or more PK parameters. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants evaluable at specified time-points. As planned, this outcome measure was analyzed in Phase 1 only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 4 | 4 | 7 | 6 | 6 | 6 | 7 | 7 | 7 | 8 | 5
nanograms per milliliter (ng/mL)
  Cycle 1 Day 1 | 14.0 (74.6) | 22.5 (19.7) | 46.1 (45.3) | 61.0 (69.0) | 124 (80.9) | 314 (37.8) | 417 (33.4) | 446 (27.4) | 738 (37.1) | 685 (30.4) | 773 (49.3) | 887 (54.5) | 668 (32.9) | 1410 (46.8) | 1100 (36.4)
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 2 | 4 | 3 | 3 | 4 | 6 | 5 | 5 | 6 | 6 | 6 | 6 | 6 | 5
  Cycle 1 Day 8 |  | 22.5 (22.8) | 33.8 (35.7) | 114 (103.6) | 108 (39.2) | 428 (49.9) | 343 (26.6) | 405 (35.6) | 846 (33.3) | 923 (69.0) | 654 (57.5) | 852 (66.2) | 653 (69.6) | 1460 (65.7) | 825 (22.3)

7. Secondary Outcome: Phase 1, Tmax: Time to Reach the Maximum Observed Plasma Concentration (Cmax) for TAK-981
Description: Tmax for TAK-981 was reported.
Time Frame: as for outcome 6
Population: PK analysis set consisted of participants with sufficient dosing and PK data to reliably estimate 1 or more PK parameters. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants evaluable at specified time-points. As planned, this outcome measure was analyzed in Phase 1 only.
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 4 | 4 | 7 | 6 | 6 | 6 | 7 | 7 | 7 | 8 | 5
hours
  Cycle 1 Day 1 | 1.17 [1.08 to 1.62] | 1.22 [1.03 to 1.33] | 1.03 [0.93 to 1.08] | 1.08 [1.07 to 1.65] | 1.08 [1.07 to 1.57] | 1.18 [1.05 to 2.13] | 1.12 [1.00 to 1.68] | 1.08 [1.00 to 1.40] | 1.02 [0.97 to 1.20] | 1.17 [1.08 to 1.22] | 1.03 [1.00 to 1.13] | 1.12 [1.05 to 1.25] | 1.17 [1.03 to 1.25] | 1.11 [1.07 to 1.27] | 1.05 [1.02 to 1.17]
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 2 | 4 | 3 | 3 | 4 | 6 | 5 | 5 | 6 | 6 | 6 | 6 | 6 | 5
  Cycle 1 Day 8 |  | 1.19 [1.13 to 1.25] | 1.17 [1.07 to 2.08] | 1.03 [1.00 to 1.05] | 1.10 [1.03 to 1.42] | 1.09 [1.00 to 1.23] | 1.09 [1.03 to 1.13] | 1.13 [1.00 to 1.25] | 1.05 [1.00 to 1.17] | 1.05 [0.95 to 1.35] | 1.03 [1.00 to 1.12] | 1.12 [1.10 to 1.75] | 1.15 [0.98 to 3.08] | 1.08 [1.00 to 1.22] | 1.13 [1.08 to 1.17]

8. Secondary Outcome: Phase 1, AUC0-last: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-981
Description: AUC0-last for TAK-981 was reported.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms per milliliter (h*ng/mL)
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 4 | 4 | 7 | 6 | 6 | 6 | 7 | 7 | 7 | 8 | 5
hours*nanograms per milliliter (h*ng/mL)
  Cycle 1 Day 1 | 50.1 (35.0) | 98.4 (15.5) | 178 (19.6) | 289 (40.6) | 438 (34.5) | 939 (20.7) | 1070 (28.2) | 1020 (25.8) | 1310 (16.9) | 1330 (15.7) | 1460 (31.0) | 1670 (31.9) | 1410 (31.8) | 2510 (30.1) | 1890 (39.7)
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 2 | 4 | 3 | 3 | 4 | 6 | 5 | 5 | 6 | 6 | 6 | 6 | 6 | 5
  Cycle 1 Day 8 |  | 98.6 (13.5) | 174 (23.0) | 364 (58.0) | 405 (20.3) | 1020 (31.1) | 906 (30.6) | 931 (19.5) | 1220 (19.1) | 1310 (33.0) | 1230 (31.1) | 1650 (47.6) | 1300 (59.2) | 3050 (81.2) | 1620 (23.4)

9. Secondary Outcome: Phase 1, AUC0-inf: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-981
Description: AUC0-inf for TAK-981 was reported.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 4 | 4 | 7 | 6 | 6 | 6 | 7 | 7 | 6 | 7 | 5
h*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 3 | 4 | 3 | 4 | 4 | 7 | 6 | 6 | 6 | 7 | 7 | 6 | 7 | 3
  Cycle 1 Day 1 | 53.5 (31.1) | 100 (14.7) | 181 (19.5) | 294 (39.2) | 443 (34.7) | 949 (20.2) | 1090 (28.0) | 1040 (26.1) | 1330 (17.0) | 1350 (15.5) | 1480 (31.6) | 1700 (31.7) | 1360 (32.3) | 2540 (33.3) | 2280 (5.6)
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 2 | 4 | 3 | 3 | 4 | 5 | 5 | 4 | 6 | 6 | 6 | 5 | 5 | 5
  Cycle 1 Day 8 |  | 103 (12.8) | 183 (21.9) | 382 (53.5) | 438 (16.2) | 1050 (29.9) | 897 (30.7) | 967 (20.6) | 1260 (21.9) | 1410 (31.4) | 1310 (28.3) | 1710 (46.8) | 1190 (40.8) | 2590 (60.2) | 1710 (24.4)

10. Secondary Outcome: Phase 1, t1/2z: Terminal Disposition Phase Half-life for TAK-981
Description: t1/2z for TAK-981 was reported.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 4 | 4 | 7 | 6 | 6 | 6 | 7 | 7 | 6 | 7 | 5
hours
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 3 | 4 | 3 | 4 | 4 | 7 | 6 | 6 | 6 | 7 | 7 | 6 | 7 | 3
  Cycle 1 Day 1 | 5.41 [2.92 to 6.40] | 7.37 [4.90 to 9.90] | 7.60 [6.92 to 8.49] | 7.88 [5.81 to 10.32] | 7.87 [7.30 to 9.78] | 8.12 [6.77 to 9.19] | 9.18 [8.05 to 10.95] | 8.89 [6.56 to 11.81] | 9.44 [7.58 to 10.23] | 9.62 [7.30 to 10.48] | 8.01 [5.39 to 9.90] | 8.32 [7.06 to 13.77] | 8.38 [7.01 to 10.74] | 8.99 [7.38 to 11.67] | 8.61 [7.01 to 9.74]
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 2 | 4 | 3 | 3 | 4 | 5 | 5 | 4 | 6 | 6 | 6 | 5 | 5 | 5
  Cycle 1 Day 8 |  | 5.74 [5.65 to 5.83] | 6.02 [4.53 to 6.74] | 6.08 [4.51 to 7.45] | 6.38 [6.12 to 10.33] | 5.73 [5.03 to 6.14] | 6.47 [5.15 to 6.59] | 6.16 [5.26 to 7.36] | 4.64 [3.12 to 6.81] | 2.95 [2.32 to 7.30] | 5.45 [3.02 to 6.13] | 6.54 [5.40 to 7.02] | 5.43 [3.00 to 6.20] | 6.20 [6.03 to 16.02] | 6.36 [3.12 to 7.16]

11. Secondary Outcome: Phase 1, CL: Total Clearance for TAK-981
Description: CL for TAK-981 was reported.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 4 | 4 | 7 | 6 | 6 | 6 | 7 | 7 | 6 | 7 | 5
liter per hour (L/h)
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 3 | 4 | 3 | 4 | 4 | 7 | 6 | 6 | 6 | 7 | 7 | 6 | 7 | 3
  Cycle 1 Day 1 | 56.1 (31.1) | 59.8 (14.7) | 55.3 (19.5) | 51.0 (39.2) | 56.4 (34.7) | 42.2 (20.2) | 55.3 (28.0) | 57.8 (26.1) | 56.3 (17.0) | 55.7 (15.5) | 60.7 (31.6) | 52.9 (31.7) | 66.0 (32.3) | 47.3 (33.3) | 52.6 (5.6)
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 2 | 4 | 3 | 3 | 4 | 5 | 5 | 4 | 6 | 6 | 6 | 5 | 5 | 5
  Cycle 1 Day 8 |  | 58.3 (12.8) | 54.7 (21.9) | 39.3 (53.5) | 57.1 (16.2) | 38.1 (29.9) | 66.9 (30.7) | 62.0 (20.6) | 59.4 (21.9) | 53.1 (31.4) | 68.8 (28.3) | 52.8 (46.8) | 75.6 (40.8) | 46.4 (60.2) | 70.3 (24.4)

12. Secondary Outcome: Phase 1, Vss: Volume of Distribution at Steady State for TAK-981
Description: Vss for TAK-981 was reported.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 4 | 4 | 7 | 6 | 6 | 6 | 7 | 7 | 6 | 7 | 5
liters
  Cycle 1 Day 1: number analyzed (Participants) | 5 | 3 | 4 | 3 | 4 | 4 | 7 | 6 | 6 | 6 | 7 | 7 | 6 | 7 | 3
  Cycle 1 Day 1 | 332 (37.9) | 437 (18.2) | 443 (28.9) | 411 (72.8) | 392 (39.9) | 234 (36.0) | 359 (33.5) | 367 (19.2) | 311 (24.0) | 345 (29.1) | 314 (46.3) | 290 (59.4) | 396 (25.8) | 271 (31.3) | 288 (27.6)
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 2 | 4 | 3 | 3 | 4 | 5 | 5 | 4 | 6 | 6 | 6 | 5 | 5 | 5
  Cycle 1 Day 8 |  | 385 (12.9) | 390 (32.0) | 233 (119.7) | 441 (41.0) | 173 (51.7) | 400 (32.2) | 334 (21.2) | 185 (48.8) | 144 (84.8) | 285 (39.3) | 241 (76.2) | 307 (60.6) | 255 (36.6) | 322 (32.7)

13. Secondary Outcome: Phase 1: ORR
Description: ORR was defined as percentage of participants who achieved CR or PR during the study as determined by the investigator according to response assessments based on RECIST v1.1 for solid tumors or Lugano classification for lymphoma.
Time Frame: From the first dose of study drug until first PD or death, whichever occurred first (up to 34.3 months)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 4 | 3 | 6 | 6 | 6 | 6 | 7 | 6 | 5 | 7 | 5
percentage of participants | 0.0 [0.00 to 60.24] | 0.0 [0.00 to 70.76] | 0.0 [0.00 to 60.24] | 0.0 [0.00 to 70.76] | 0.0 [0.00 to 60.24] | 33.3 [0.84 to 90.57] | 0.0 [0.00 to 45.93] | 0.0 [0.00 to 45.93] | 0.0 [0.0 to 45.93] | 0.0 [0.0 to 45.93] | 0.0 [0.0 to 40.96] | 16.7 [0.42 to 64.12] | 0.0 [0.0 to 52.18] | 14.3 [0.36 to 57.87] | 0.0 [0.00 to 52.18]

14. Secondary Outcome: Phase 1 and 2: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants who achieved stable disease (SD) (greater than [>] 6 weeks) or better as determined by the investigator according to RECIST v1.1 for solid tumors or Lugano classification for lymphoma.
Time Frame: From first dose of study drug up to 34.3 months (for Phase 1) and up to 11.2 months (for Phase 2)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW | Phase 2, Dose Expansion, Cohort A, NSCLC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort B, Cervical Cancer: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort C, MSS-CRC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort D, DLBCL After CAR T-cells Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort E, DLBCL Without Prior Cellular Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort F, Follicular Lymphoma: TAK-981 90 mg BIW
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 4 | 3 | 6 | 6 | 6 | 6 | 7 | 6 | 5 | 7 | 5 | 7 | 3 | 6 | 4 | 3 | 1
percentage of participants | 0.0 [0.0 to 60.24] | 0.0 [0.0 to 70.76] | 25.0 [0.63 to 80.59] | 33.3 [0.84 to 90.57] | 75.0 [19.41 to 99.37] | 66.7 [9.43 to 99.16] | 0.0 [0.0 to 45.93] | 66.7 [22.28 to 95.67] | 16.7 [0.42 to 64.12] | 66.7 [22.28 to 95.67] | 42.9 [9.90 to 81.59] | 50.0 [11.81 to 88.19] | 60.0 [14.66 to 94.73] | 42.9 [9.90 to 81.59] | 20.0 [0.51 to 71.64] | 71.4 [29.04 to 96.33] | 66.7 [9.43 to 99.16] | 33.3 [4.33 to 77.72] | 0.0 [0.0 to 60.24] | 0.0 [0.00 to 70.76] | 100.0 [2.50 to 100.0]

15. Secondary Outcome: Phase 1 and 2: Duration of Response (DOR)
Description: DOR was defined as the time from the date of first documentation of a PR or better to the date of first documentation of PD for responders (PR or better) and determined by the investigator according to RECIST v1.1 with solid tumors or Lugano classification for lymphoma.
Time Frame: From first documented confirmed CR or PR until first documentation of PD up to 34.3 months (for Phase 1) and up to 11.2 months (for Phase 2)
Population: Tumor response-evaluable analysis set consisted of participants who received at least 1 dose of study drug, had sites of measurable disease at baseline, and 1 postbaseline disease assessment, or was discontinued due to symptomatic deterioration or death before a postbaseline evaluation happened. Here, "overall number of participants analyzed" signifies participants who had CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW | Phase 2, Dose Expansion, Cohort A, NSCLC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort B, Cervical Cancer: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort C, MSS-CRC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort D, DLBCL After CAR T-cells Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort E, DLBCL Without Prior Cellular Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort F, Follicular Lymphoma: TAK-981 90 mg BIW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
months |  |  |  |  |  | 6.93 [NA to NA] — Upper and lower limit of 95% confidence internal (CI) could not be estimated due to insufficient number of participants with events. |  |  |  |  |  | 1.41 [NA to NA] — Upper and lower limit of 95% CI could not be estimated due to insufficient number of participants with events. |  | NA [NA to NA] — Median, upper and lower limit of 95% CI could not be estimated due to insufficient number of participants with events. |  |  |  |  |  |  | 5.55 [NA to NA] — Upper and lower limit of 95% CI could not be estimated due to insufficient number of participants with events.

16. Secondary Outcome: Phase 1 and 2: Time to Progression (TTP)
Description: TTP was defined as the time from the date of the first dose administration to the date of first documented PD as determined by the investigator according to RECIST v1.1 for solid tumors or Lugano classification for lymphoma.
Time Frame: From first dose of study drug to the date of the first documentation of PD up to 34.3 months (for Phase 1) and up to 11.2 months (for Phase 2)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW | Phase 2, Dose Expansion, Cohort A, NSCLC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort B, Cervical Cancer: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort C, MSS-CRC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort D, DLBCL After CAR T-cells Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort E, DLBCL Without Prior Cellular Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort F, Follicular Lymphoma: TAK-981 90 mg BIW
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 4 | 4 | 7 | 6 | 6 | 6 | 8 | 7 | 7 | 8 | 6 | 7 | 3 | 7 | 4 | 3 | 1
months | 1.18 [0.72 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 0.79 [0.76 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 1.38 [0.59 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 1.25 [1.18 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 2.10 [1.38 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 5.49 [1.25 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 1.21 [0.46 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 3.75 [0.72 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 1.28 [1.22 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 2.71 [1.35 to 8.08] | 6.97 [2.66 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 3.94 [1.18 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 2.79 [1.25 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [1.38 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 1.97 [1.74 to 2.04] | 6.06 [2.07 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 3.78 [0.99 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 1.18 [0.92 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 1.04 [0.59 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 1.09 [0.43 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 11.17 [NA to NA] — Upper and lower limit of 95% CI could not be estimated due to insufficient number of participants with events.

17. Secondary Outcome: Phase 1 and 2: Time to Response (TTR)
Description: TTR was defined as the time from the date of first study drug administration to the date of first documented PR or better by the investigator for responders according to RECIST v1.1 for solid tumors or Lugano classification for lymphoma. Here, "overall number of participants analyzed" signifies participants who had CR or PR.
Time Frame: From first dose of study drug to the date of the first documentation of PR or better, whichever occurred first up to 34.3 months (for Phase 1) and up to 11.2 months (for Phase 2)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW | Phase 2, Dose Expansion, Cohort A, NSCLC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort B, Cervical Cancer: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort C, MSS-CRC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort D, DLBCL After CAR T-cells Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort E, DLBCL Without Prior Cellular Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort F, Follicular Lymphoma: TAK-981 90 mg BIW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
months |  |  |  |  |  | NA [1.38 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. |  |  |  |  |  | NA [3.91 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. |  | NA [1.74 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. |  |  |  |  |  |  | 5.65 [NA to NA] — Upper limit and lower limit of 95% CI could not be estimated due to insufficient number of participants with events.

18. Secondary Outcome: Phase 1 and 2: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of the first dose administration to the date of first documentation of PD or death due to any cause, whichever occurs first as determined by the investigator according to RECIST v1.1 for solid tumors or Lugano classification for lymphoma.
Time Frame: From the first dose of study drug to date of PD or death, whichever occurred first up to 34.3 months (for Phase 1) and up to 11.2 months (for Phase 2)
Population: Safety analysis set consisted of participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW | Phase 2, Dose Expansion, Cohort A, NSCLC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort B, Cervical Cancer: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort C, MSS-CRC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort D, DLBCL After CAR T-cells Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort E, DLBCL Without Prior Cellular Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort F, Follicular Lymphoma: TAK-981 90 mg BIW
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 4 | 4 | 7 | 6 | 6 | 6 | 8 | 7 | 7 | 8 | 6 | 7 | 3 | 7 | 4 | 3 | 1
months | 0.95 [0.46 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 0.79 [0.76 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 1.38 [0.59 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 1.25 [1.18 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 2.10 [1.38 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 5.49 [1.25 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 1.18 [0.46 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 2.53 [1.02 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 1.27 [1.22 to 1.54] | 2.71 [1.35 to 8.08] | 2.66 [0.82 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 3.94 [1.18 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 2.79 [1.25 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 3.32 [1.38 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 1.97 [1.74 to 2.04] | 6.06 [2.07 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 3.78 [0.99 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 1.18 [0.92 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 1.38 [0.59 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 1.09 [0.43 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 11.17 [NA to NA] — Upper limit and lower limit of 95% CI could not be estimated due to insufficient number of participants with events.

19. Secondary Outcome: Phase 1 and 2: Overall Survival (OS)
Description: OS was defined as the time from the date of the first dose administration to the date of death.
Time Frame: From date of first dose of study drug up to death up to 34.3 months (for Phase 1) and up to 11.2 months (for Phase 2)
Population: Safety analysis set consisted of participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW | Phase 2, Dose Expansion, Cohort A, NSCLC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort B, Cervical Cancer: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort C, MSS-CRC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort D, DLBCL After CAR T-cells Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort E, DLBCL Without Prior Cellular Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort F, Follicular Lymphoma: TAK-981 90 mg BIW
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 4 | 4 | 7 | 6 | 6 | 6 | 8 | 7 | 7 | 8 | 6 | 7 | 3 | 7 | 4 | 3 | 1
months | NA [0.46 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [NA to NA] — Median, upper limit and lower limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [NA to NA] — Median, upper limit and lower limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [NA to NA] — Median, upper limit and lower limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [3.02 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [1.48 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [1.25 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [NA to NA] — Median, upper limit and lower limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [NA to NA] — Median, upper limit and lower limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [NA to NA] — Median, upper limit and lower limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [0.82 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 5.49 [5.49 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [1.77 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [5.22 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [NA to NA] — Median, upper limit and lower limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [1.87 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [3.29 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [1.87 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 2.43 [1.28 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 6.14 [1.58 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [NA to NA] — Median, upper limit and lower limit of 95% CI could not be estimated due to insufficient number of participants with events.

20. Secondary Outcome: Phase 1: Fold Change From Baseline in Levels of TAK-981 Small Ubiquitin-like Modifier (SUMO) Adduct Formation in Blood Lymphocytes
Description: TAK-981-SUMO adduct formation in peripheral blood lymphocytes was tested by flow cytometry with an antibody recognizing the TAK-981-SUMO adduct formation during the inhibition of the SUMO-activating enzyme by TAK-981.
Time Frame: Cycle 1 Day 1: 1, 4 and 8 hours post-dose; Cycle 1 Day 8: Pre-dose, 1, 4 and 8 hours post-dose (Cycle length = 21 days)
Population: Pharmacodynamic analysis set consisted of participants who provided evaluable blood samples (Cycle 1 Day 1 pre-dose sample and at least 1 post-dose sample). Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and here, "number analyzed" signifies participants evaluable at specified time-points.
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 4 | 7 | 6 | 6 | 6 | 8 | 7 | 7 | 8 | 6
fold change
  Cycle 1 Day 1: 1 hour post-dose: number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 4 | 7 | 6 | 6 | 6 | 8 | 7 | 7 | 8 | 6
  Cycle 1 Day 1: 1 hour post-dose | 1.8 (0.21) | 2.3 (0.16) | 2.9 (1.38) | 5.9 (0.83) | 5.9 (1.07) | 8.4 (1.25) | 7.5 (2.57) | 6.5 (2.27) | 7.8 (1.59) | 7.0 (2.03) | 8.5 (1.10) | 8.8 (1.46) | 8.1 (2.12) | 8.5 (2.12) | 8.1 (1.41)
  Cycle 1 Day 1: 4 hour post-dose | 1.6 (0.19) | 2.1 (0.04) | 2.6 (1.64) | 4.8 (0.70) | 5.1 (0.74) | 5.8 (0.44) | 6.2 (2.15) | 4.7 (1.57) | 5.8 (0.86) | 5.8 (1.05) | 6.0 (1.05) | 6.2 (1.10) | 5.9 (1.42) | 6.2 (1.32) | 5.8 (1.22)
  Cycle 1 Day 1: 8 hour post-dose: number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 4 | 7 | 5 | 6 | 6 | 8 | 7 | 7 | 8 | 6
  Cycle 1 Day 1: 8 hour post-dose | 1.5 (0.23) | 1.9 (0.08) | 2.7 (1.36) | 4.3 (0.85) | 4.6 (0.77) | 4.9 (0.10) | 4.3 (2.05) | 3.3 (1.02) | 5.2 (1.49) | 4.8 (1.10) | 4.7 (1.02) | 5.5 (1.32) | 4.9 (1.20) | 5.0 (0.94) | 4.0 (1.21)
  Cycle 1 Day 8: Pre-dose: number analyzed (Participants) | 0 | 2 | 4 | 3 | 3 | 4 | 7 | 5 | 6 | 6 | 6 | 6 | 7 | 5 | 4
  Cycle 1 Day 8: Pre-dose |  | 1.8 (0.27) | 2.0 (0.80) | 3.6 (0.92) | 3.3 (0.31) | 2.9 (0.87) | 2.9 (1.20) | 2.1 (0.30) | 3.9 (0.75) | 2.1 (0.66) | 2.6 (0.92) | 2.4 (0.53) | 2.4 (0.62) | 3.7 (1.06) | 2.3 (0.38)
  Cycle 1 Day 8: 1 hour post-dose: number analyzed (Participants) | 0 | 2 | 4 | 3 | 3 | 4 | 6 | 5 | 6 | 6 | 6 | 6 | 7 | 4 | 4
  Cycle 1 Day 8: 1 hour post-dose |  | 3.2 (0.72) | 3.8 (1.73) | 8.0 (3.03) | 7.9 (2.00) | 8.4 (2.20) | 9.6 (3.94) | 6.9 (0.89) | 8.7 (2.91) | 7.4 (2.95) | 7.5 (2.18) | 9.6 (1.74) | 8.4 (2.68) | 9.2 (1.79) | 8.2 (1.94)
  Cycle 1 Day 8: 4 hour post-dose: number analyzed (Participants) | 0 | 2 | 4 | 3 | 3 | 4 | 6 | 5 | 6 | 6 | 6 | 6 | 7 | 4 | 5
  Cycle 1 Day 8: 4 hour post-dose |  | 2.9 (0.62) | 3.4 (1.55) | 7.1 (2.38) | 7.2 (1.84) | 6.3 (2.01) | 7.3 (3.17) | 5.3 (0.55) | 7.1 (1.47) | 5.9 (2.37) | 6.9 (0.85) | 6.9 (1.58) | 6.2 (1.81) | 7.9 (1.90) | 6.1 (1.30)
  Cycle 1 Day 8: 8 hour post-dose: number analyzed (Participants) | 0 | 2 | 4 | 3 | 3 | 4 | 6 | 4 | 6 | 6 | 6 | 6 | 6 | 4 | 5
  Cycle 1 Day 8: 8 hour post-dose |  | 2.9 (0.65) | 3.2 (1.53) | 6.7 (1.98) | 6.0 (1.42) | 6.1 (2.45) | 6.3 (2.63) | 4.3 (0.59) | 6.6 (1.68) | 5.2 (2.05) | 5.8 (1.19) | 5.7 (1.05) | 5.8 (2.04) | 5.9 (0.83) | 5.2 (1.06)

21. Secondary Outcome: Phase 1: Fold Change From Baseline in Levels of TAK-981 SUMO Adduct Formation in Skin
Description: TAK-981-SUMO adduct formation in skin was tested by flow cytometry with an antibody recognizing the TAK-981-SUMO adduct formation during the inhibition of the SUMO-activating enzyme by TAK-981.
Time Frame: Cycle 1 Day 8 (Cycle length = 21 days)
Population: Pharmacodynamic analysis set consisted of participants who provided evaluable skin biopsies (screening sample and at least 1 on-treatment sample). Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
fold change |  |  | 115.57 (NA) — Standard Deviation could not be estimated due to insufficient number of participants available for analysis. |  |  |  |  |  |  |  |  | 1343.23 (NA) — Standard Deviation could not be estimated due to insufficient number of participants available for analysis. |  |  |

22. Secondary Outcome: Phase 1: Fold Change From Baseline in SUMO Pathway Inhibition in Blood Lymphocytes
Description: SUMO pathway inhibition in peripheral blood lymphocytes was tested by flow cytometry with an antibody recognizing SUMO-2/3 chains.
Time Frame: Cycle 1 Day 1: 1, 4 and 8 hours post-dose; Cycle 1 Day 8: Pre-dose, 1, 4 and 8 hours post-dose (Cycle length = 21 days)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 4 | 7 | 6 | 6 | 6 | 8 | 7 | 7 | 8 | 6
fold change
  Cycle 1 Day 1: 1 hour post-dose: number analyzed (Participants) | 3 | 3 | 4 | 3 | 3 | 4 | 7 | 6 | 6 | 6 | 8 | 7 | 7 | 8 | 6
  Cycle 1 Day 1: 1 hour post-dose | 1.0 (0.04) | 1.0 (0.05) | 0.9 (0.11) | 0.9 (0.04) | 0.9 (0.06) | 4.7 (7.88) | 0.8 (0.13) | 0.7 (0.13) | 0.6 (0.14) | 0.6 (0.11) | 0.6 (0.11) | 0.6 (0.12) | 0.6 (0.09) | 0.5 (0.07) | 0.6 (0.22)
  Cycle 1 Day 1: 4 hour post-dose | 0.9 (0.15) | 1.0 (0.07) | 1.0 (0.07) | 0.9 (0.05) | 1.0 (0.09) | 4.1 (6.38) | 2.3 (4.03) | 0.9 (0.41) | 0.5 (0.20) | 2.5 (4.74) | 0.6 (0.13) | 0.6 (0.18) | 0.6 (0.11) | 0.5 (0.14) | 0.6 (0.36)
  Cycle 1 Day 1: 8 hour post-dose: number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 4 | 7 | 5 | 6 | 6 | 8 | 7 | 7 | 8 | 6
  Cycle 1 Day 1: 8 hour post-dose | 1.0 (0.20) | 1.0 (0.12) | 1.0 (0.19) | 1.0 (0.07) | 0.9 (0.18) | 4.0 (6.19) | 0.7 (0.18) | 0.7 (0.25) | 0.6 (0.26) | 2.5 (4.49) | 0.6 (0.17) | 0.7 (0.13) | 0.6 (0.11) | 0.6 (0.23) | 0.6 (0.35)
  Cycle 1 Day 8: Pre-dose: number analyzed (Participants) | 0 | 2 | 4 | 3 | 3 | 4 | 7 | 5 | 6 | 6 | 6 | 6 | 7 | 5 | 4
  Cycle 1 Day 8: Pre-dose |  | 1.0 (0.17) | 1.0 (0.15) | 1.1 (0.16) | 1.7 (0.82) | 5.5 (9.42) | 2.1 (3.57) | 1.5 (0.66) | 1.0 (0.24) | 1.0 (0.16) | 0.8 (0.43) | 1.1 (0.27) | 1.0 (0.18) | 1.1 (0.21) | 2.8 (3.74)
  Cycle 1 Day 8: 1 hour post-dose: number analyzed (Participants) | 0 | 2 | 4 | 3 | 3 | 4 | 6 | 5 | 6 | 6 | 6 | 6 | 7 | 4 | 4
  Cycle 1 Day 8: 1 hour post-dose |  | 1.0 (0.16) | 1.0 (0.14) | 0.9 (0.10) | 1.6 (0.68) | 4.6 (8.08) | 0.6 (0.35) | 0.9 (0.41) | 0.5 (0.24) | 0.6 (0.22) | 0.5 (0.23) | 0.7 (0.19) | 0.5 (0.09) | 0.6 (0.17) | 1.5 (2.00)
  Cycle 1 Day 8: 4 hour post-dose: number analyzed (Participants) | 0 | 2 | 4 | 3 | 3 | 4 | 6 | 5 | 6 | 6 | 6 | 6 | 7 | 4 | 5
  Cycle 1 Day 8: 4 hour post-dose |  | 1.0 (0.15) | 1.0 (0.15) | 1.0 (0.08) | 1.7 (0.77) | 4.6 (7.98) | 0.7 (0.31) | 1.0 (0.51) | 0.6 (0.22) | 1.8 (3.05) | 0.7 (0.16) | 0.7 (0.19) | 0.6 (0.14) | 0.7 (0.19) | 1.5 (1.87)
  Cycle 1 Day 8: 8 hour post-dose: number analyzed (Participants) | 0 | 2 | 4 | 3 | 3 | 4 | 6 | 4 | 6 | 6 | 6 | 6 | 6 | 4 | 5
  Cycle 1 Day 8: 8 hour post-dose |  | 1.1 (0.10) | 1.0 (0.23) | 0.9 (0.11) | 1.7 (0.65) | 4.6 (8.20) | 0.7 (0.30) | 1.0 (0.76) | 0.6 (0.18) | 1.9 (3.06) | 0.8 (0.19) | 0.7 (0.20) | 0.6 (0.21) | 0.6 (0.18) | 1.5 (2.14)

23. Secondary Outcome: Phase 1: Fold Change From Baseline in SUMO Pathway Inhibition in Skin
Description: SUMO pathway inhibition in skin was tested by flow cytometry with an antibody recognizing SUMO-2/3 chains.
Time Frame: Cycle 1 Day 8 (Cycle length = 21 days)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 4 | 4 | 5 | 5 | 6 | 6 | 6 | 6 | 6 | 6 | 6
fold change | 1.01 (0.067) | 0.71 (0.398) | 0.82 (0.088) | 0.91 (0.233) | 1.05 (0.122) | 0.86 (0.146) | 0.72 (0.276) | 0.73 (0.298) | 0.64 (0.156) | 0.71 (0.224) | 0.56 (0.136) | 0.65 (0.298) | 0.78 (0.123) | 0.42 (0.376) | 0.44 (0.210)

24. Secondary Outcome: Phase 2: Number of Participants Reporting One or More TEAEs
Description: TEAEs were AEs that occurred after administration of the first dose of any study drug and through 30 days after the last dose of any study drug. AE means any untoward medical occurrence in a participant administered a pharmaceutical product. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product. Any abnormal laboratory results were reported as TEAEs.
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (up to 12.2 months)
Population: Safety analysis set consisted of participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2, Dose Expansion, Cohort A, NSCLC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort B, Cervical Cancer: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort C, MSS-CRC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort D, DLBCL After CAR T-cells Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort E, DLBCL Without Prior Cellular Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort F, Follicular Lymphoma: TAK-981 90 mg BIW
Number analyzed (Participants) | 7 | 3 | 7 | 4 | 3 | 1
Participants | 6 | 3 | 7 | 4 | 3 | 1

25. Secondary Outcome: Phase 2: Number of Participants With Grade 3 or Higher TEAEs
Description: The severity grade was evaluated as per the CTCAE Version 5.0, except for CRS, which was assessed by ASTCT consensus grading. Where Grade 3 was severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL, Grade 4 was 4 Life-threatening consequences; urgent intervention indicated. and Grade 5 was death related to AE. TEAEs were AEs that occurred after administration of the first dose of any study drug and through 30 days after the last dose of any study drug.
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (up to 12.2 months)
Population: Safety analysis set consisted of participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2, Dose Expansion, Cohort A, NSCLC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort B, Cervical Cancer: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort C, MSS-CRC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort D, DLBCL After CAR T-cells Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort E, DLBCL Without Prior Cellular Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort F, Follicular Lymphoma: TAK-981 90 mg BIW
Number analyzed (Participants) | 7 | 3 | 7 | 4 | 3 | 1
Participants | 4 | 1 | 6 | 3 | 3 | 1

26. Secondary Outcome: Phase 2: Duration of TEAEs
Description: as for outcome 3
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (up to 12.2 months)
Population: Safety analysis set consisted of participants who received at least 1 dose, even if incomplete, of study drug.
Measure: Median (Full Range); unit: days
Arm/Group | Phase 2, Dose Expansion, Cohort A, NSCLC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort B, Cervical Cancer: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort C, MSS-CRC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort D, DLBCL After CAR T-cells Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort E, DLBCL Without Prior Cellular Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort F, Follicular Lymphoma: TAK-981 90 mg BIW
Number analyzed (Participants) | 7 | 3 | 7 | 4 | 3 | 1
days | 8.5 [1 to 336] | 4.0 [1 to 45] | 5.0 [1 to 72] | 5.0 [1 to 26] | 3.0 [1 to 19] | 1.0 [1 to 56]

ADVERSE EVENTS:
Time Frame: Serious and Other (Non-serious) AEs: From the first dose of study drug through 30 days after the last dose of study drug up to 35.3 months (for Phase 1) and up to 12.2 months (for Phase 2); All-cause mortality: From date of first dose of study drug up to death due to any cause (up to 34.3 months for Phase 1 and up to 11.2 months for Phase 2)
Arm/Group | Phase 1, Dose Escalation: TAK-981 3 mg BIW | Phase 1, Dose Escalation: TAK-981 6 mg BIW | Phase 1, Dose Escalation: TAK-981 10 mg BIW | Phase 1, Dose Escalation: TAK-981 15 mg BIW | Phase 1, Dose Escalation: TAK-981 25 mg BIW | Phase 1, Dose Escalation: TAK-981 40 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg BIW | Phase 1, Dose Escalation: TAK-981 60 mg QW | Phase 1, Dose Escalation: TAK-981 75 mg BIW | Phase 1, Dose Escalation: TAK-981 75 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg BIW | Phase 1, Dose Escalation: TAK-981 90 mg QW | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 | Phase 1, Dose Escalation: TAK-981 120 mg BIW | Phase 1, Dose Escalation: TAK-981 120 mg QW | Phase 2, Dose Expansion, Cohort A, NSCLC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort B, Cervical Cancer: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort C, MSS-CRC: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort D, DLBCL After CAR T-cells Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort E, DLBCL Without Prior Cellular Therapy: TAK-981 90 mg BIW | Phase 2, Dose Expansion, Cohort F, Follicular Lymphoma: TAK-981 90 mg BIW
All-Cause Mortality (participants affected / at risk) | 1/5 | 0/3 | 0/4 | 0/3 | 1/4 | 1/4 | 2/7 | 1/6 | 1/6 | 0/6 | 2/8 | 2/7 | 1/7 | 1/8 | 0/6 | 1/7 | 1/3 | 1/7 | 4/4 | 2/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 3/5 | 2/3 | 3/4 | 1/3 | 2/4 | 2/4 | 3/7 | 1/6 | 3/6 | 1/6 | 5/8 | 2/7 | 2/7 | 5/8 | 2/6 | 2/7 | 1/3 | 4/7 | 2/4 | 2/3 | 0/1
Other Adverse Events (participants affected / at risk) | 4/5 | 3/3 | 4/4 | 2/3 | 4/4 | 4/4 | 6/7 | 6/6 | 5/6 | 6/6 | 7/8 | 7/7 | 7/7 | 8/8 | 6/6 | 6/7 | 3/3 | 7/7 | 4/4 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1, Dose Escalation: TAK-981 3 mg BIW (N=5) | Phase 1, Dose Escalation: TAK-981 6 mg BIW (N=3) | Phase 1, Dose Escalation: TAK-981 10 mg BIW (N=4) | Phase 1, Dose Escalation: TAK-981 15 mg BIW (N=3) | Phase 1, Dose Escalation: TAK-981 25 mg BIW (N=4) | Phase 1, Dose Escalation: TAK-981 40 mg BIW (N=4) | Phase 1, Dose Escalation: TAK-981 60 mg BIW (N=7) | Phase 1, Dose Escalation: TAK-981 60 mg QW (N=6) | Phase 1, Dose Escalation: TAK-981 75 mg BIW (N=6) | Phase 1, Dose Escalation: TAK-981 75 mg QW (N=6) | Phase 1, Dose Escalation: TAK-981 90 mg BIW (N=8) | Phase 1, Dose Escalation: TAK-981 90 mg QW (N=7) | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 (N=7) | Phase 1, Dose Escalation: TAK-981 120 mg BIW (N=8) | Phase 1, Dose Escalation: TAK-981 120 mg QW (N=6) | Phase 2, Dose Expansion, Cohort A, NSCLC: TAK-981 90 mg BIW (N=7) | Phase 2, Dose Expansion, Cohort B, Cervical Cancer: TAK-981 90 mg BIW (N=3) | Phase 2, Dose Expansion, Cohort C, MSS-CRC: TAK-981 90 mg BIW (N=7) | Phase 2, Dose Expansion, Cohort D, DLBCL After CAR T-cells Therapy: TAK-981 90 mg BIW (N=4) | Phase 2, Dose Expansion, Cohort E, DLBCL Without Prior Cellular Therapy: TAK-981 90 mg BIW (N=3) | Phase 2, Dose Expansion, Cohort F, Follicular Lymphoma: TAK-981 90 mg BIW (N=1)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal mass (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1, Dose Escalation: TAK-981 3 mg BIW (N=5) | Phase 1, Dose Escalation: TAK-981 6 mg BIW (N=3) | Phase 1, Dose Escalation: TAK-981 10 mg BIW (N=4) | Phase 1, Dose Escalation: TAK-981 15 mg BIW (N=3) | Phase 1, Dose Escalation: TAK-981 25 mg BIW (N=4) | Phase 1, Dose Escalation: TAK-981 40 mg BIW (N=4) | Phase 1, Dose Escalation: TAK-981 60 mg BIW (N=7) | Phase 1, Dose Escalation: TAK-981 60 mg QW (N=6) | Phase 1, Dose Escalation: TAK-981 75 mg BIW (N=6) | Phase 1, Dose Escalation: TAK-981 75 mg QW (N=6) | Phase 1, Dose Escalation: TAK-981 90 mg BIW (N=8) | Phase 1, Dose Escalation: TAK-981 90 mg QW (N=7) | Phase 1, Dose Escalation: TAK-981 90 mg QW on Days 1, 8, 15 (N=7) | Phase 1, Dose Escalation: TAK-981 120 mg BIW (N=8) | Phase 1, Dose Escalation: TAK-981 120 mg QW (N=6) | Phase 2, Dose Expansion, Cohort A, NSCLC: TAK-981 90 mg BIW (N=7) | Phase 2, Dose Expansion, Cohort B, Cervical Cancer: TAK-981 90 mg BIW (N=3) | Phase 2, Dose Expansion, Cohort C, MSS-CRC: TAK-981 90 mg BIW (N=7) | Phase 2, Dose Expansion, Cohort D, DLBCL After CAR T-cells Therapy: TAK-981 90 mg BIW (N=4) | Phase 2, Dose Expansion, Cohort E, DLBCL Without Prior Cellular Therapy: TAK-981 90 mg BIW (N=3) | Phase 2, Dose Expansion, Cohort F, Follicular Lymphoma: TAK-981 90 mg BIW (N=1)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 3 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 4 | 2 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ammonia increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 2 | 2 | 2 | 1 | 1 | 0 | 4 | 0 | 2 | 0
Anisocoria (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 2 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood antidiuretic hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 4 | 4 | 1 | 3 | 3 | 2 | 1 | 1 | 6 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Complication associated with device (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 2 | 2 | 2 | 5 | 1 | 2 | 4 | 3 | 2 | 0 | 3 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device dislocation (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 2 | 3 | 1 | 2 | 4 | 4 | 3 | 3 | 2 | 2 | 3 | 0 | 4 | 1 | 2 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 3 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 2 | 4 | 1 | 2 | 2 | 2 | 1 | 0 | 2 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces pale (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 2 | 0 | 2 | 2 | 4 | 5 | 4 | 4 | 5 | 2 | 5 | 3 | 2 | 3 | 0 | 4 | 1 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 5 | 4 | 4 | 4 | 1 | 3 | 2 | 1 | 4 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 3 | 1 | 3 | 2 | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Infusion site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Interferon alpha level increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Interferon gamma level increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Interleukin level increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip blister (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip scab (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Middle insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 0 | 0 | 2 | 2 | 2 | 6 | 6 | 5 | 5 | 5 | 3 | 1 | 2 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 2 | 3 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ophthalmic migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic failure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Performance status decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Pleural fluid analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prothrombin level increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 3 | 3 | 4 | 2 | 2 | 6 | 3 | 2 | 1 | 5 | 1 | 1 | 1
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stoma prolapse (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary occult blood (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 4 | 3 | 4 | 4 | 3 | 0 | 0 | 1 | 1 | 0 | 0
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early due to enrollment challenges.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT03648372/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT03648372/SAP_001.pdf